CLINICAL TRIAL: NCT02549547
Title: Jump Step - A Participatory Approach to Physical Activity & Mental Wellness
Acronym: JumpStep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Foundation (Other); Mood Disorders Association of BC (Unknown); YMCA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID: H15-01932
Record Dates: First submitted 2015-09-01; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Major Depressive Disorder; Bipolar, Depression
Keywords: anxiety; depression; exercise; group; group medical visit; mood disorder; physical activity; primary care
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Anxiety Disorders; Depression; Motor Activity; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle Intervention (Experimental): Physical Activity focused, interdisciplinary, Group Medical Visits (GMVs)
  Interventions: Behavioral: Group Medical Visits

INTERVENTIONS:
Behavioral: Group Medical Visits — Cohorts will participate in a weekly series of 14 Group Medical Visits (GMVs) co-led by a psychiatrist and an exercise professional. Each two-hour Group Medical Visit will be divided into three sections:
  * Group check in/out; enter patients weekly step count into database; review and outline the day's group program - 20 minutes
  * Group discussion, regarding selected physical activity topics including psychiatric issues - 50 minutes
  * Physical activity component - 50 minutes The 'content' or curriculum of the GMVs will support participant Self-Management/Activation. Research has consistently emphasized the role of positive feedback, social support, reinforcement, goal setting, and motivation for improving person's self-perception to uptake physical activity.

SUMMARY:
The WHO, the Pan American Health Organization, the EU Council of Ministers, the World Federation of Mental Health, and the UK Royal College of Psychiatrists all agree -"there can be no health without mental health". Within Canada, 6.7M people live with a mental illness and when family and caregivers are included almost everyone is affected.

A systematic review (2014) concluded that physical activity has a significant potential for reducing depressive symptoms in people with a mental illness. Globally, physical inactivity is "pandemic". Current guidelines recommend a minimum of only a 150 minutes a week of moderately vigorous exercise but 85% of Canadians do not meet the national recommendations. How then can people with depression be motivated to become physically more active?

Group Medical Visits (GMVs) can be used to provide health services and they have proven effective in some settings, including mood disorders. As well as providing economic and resource efficiencies, the GMV model has the potential to add a 'support group/accountability' element for behavioural interventions such as physical activity promotion; such influence is not present in an individual patient-physician consultation.

"Jump Step" is a 14-week program within a GMV setting designed to motivate and support people with depression to engage in regular physical activity. The investigators seek to design, implement, and evaluate the effectiveness of the Group Medical Visits focused on promoting physical activity for patients with depression.

DETAILED DESCRIPTION:
Mental disorders, including anxiety and depression, contribute more than either cardiovascular disease or cancer to the burden of disease worldwide. Individuals with chronic diseases and major depression use more health resources, have higher degrees of functional disability, and experience higher productivity losses, compared to their counterparts without major depression. Within Canada, 6.7M people live with a mental illness and when family and caregivers are included almost everyone is affected.

A Cochrane Review examined the effectiveness of exercise in treating depression and the results of 39 trials and over 2,300 subjects confirmed a moderate effect for exercise when compared to no treatment or a control group. A smaller number of studies found no differences in efficacy between exercise and Cognitive Behavioural Therapy (CBT) and/or antidepressant therapies, the current "gold standards" for depression care. A systematic review (2014) concluded that physical activity has a significant potential for reducing depressive symptoms in people with a mental health challenge.

Globally, physical inactivity is "pandemic". Current guidelines recommend a minimum of only 150 minutes a week of moderately vigorous exercise but 85% of Canadians do not meet the national recommendations. There is no question that physical activity can be an effective treatment; how then can people dealing with depression be motivated to become physically more active?

The majority of psychiatric care for mood disorders is delivered through one-to-one consultations between a patient and psychiatrist or family physician. Treatment plans rarely include physical activity despite evidence for its effectiveness. In fact, efforts to promote physical activity within traditional clinical settings are fraught with challenges such as a lack of practitioner resources, reimbursement, time, and confidence, and poor patient retention. Instead, people are commonly prescribed powerful pharmaceuticals despite mounting evidence that these drugs should be reserved for the most serious cases of anxiety and depression. While drugs have their place, this place is firmly behind interventions such as psychotherapy and physical activity in the majority of cases of depression.

Novel strategies are needed for promoting physical activity and self-management that are also physically, financially, and psychologically accessible. Group Medical Visits (GMVs) are a promising approach to mental health care. Group Medical Visits are organized around a group of people living with a specific condition. The structure and formats of GMVs vary. Typically, in lieu of a short individual visit, a patient will participate in a longer (60-120 minutes) group visit with six to 14 other patients, led by a physician and/or other healthcare practitioner.

GMVs have been scientifically tested in an array of primary care settings over the last 10 to 15 years, including mental health[6-8]; no studies to date, though, have focused exclusively on physical activity promotion. Briefly, the theoretical rationale for this approach is a multifactorial "interdisciplinary model", including medication/treatment monitoring, patient education, social support, goal setting, and motivation for improving person's self-perception to uptake physical activity.

Within British Columbia, the Mood Disorders Association of BC has taken a leadership role in integrating Group Medical Visits into psychiatric care. Based on the success of MDABC's adult Group Medical Visits, UBC researchers collaborated with MDABC to design and prototype "Step-by-Step (SBS)." SBS was a series of 14 weekly Group Appointments designed to help patients with anxiety and/or depression incorporate physical activity as part of their treatment plan.

Co-led by a psychiatrist and an exercise therapist, each two-hour GMV combined specific participants' self-management and activation. A physical activity section in each Group Appointment provided participants instruction in techniques/exercises that they could employ in their everyday lives to become more physically active without having to attend special classes, set aside time, or make concerted efforts to "exercise".

After three months post-SBS intervention, median depression scales (PHQ-9) decreased 38% from 16 to 10 (p<0.01; IQR: 8/12); and, median anxiety scales (GAD-7) decreased 50% from 13 to 6.5 (p<0.05; IQR: 8.5/9). Median daily "steps" increased 71% from 3,366 to 5,746 (IQR: 2,610/6,237), though this was not significant (p>0.10). These data compare favourably with other interventions such as psychotherapy and medications. Fourteen of 15 participants (93.3%) completed the 14-week program and loved it!

In the design and realization of Step-by-Step the investigators intentionally 'meet participants where they were at." The intervention was not static but a dynamic constantly evolving process whereby the investigators continuously refined the program based on weekly feedback. As a result, the investigators were able to better able to meet the needs of participants though it did mean what the investigators were testing changed over the course of the intervention.

Equally, the investigators intended the program to address participants holistically, which therefore demanded a multifactorial approach. Instead of testing a single variable the investigators were examining the impact of a collection of elements as a whole. Exit interviews with participants suggested a number of factors might have led to program retention and the improvements in physical activity, depression, and anxiety. The investigators cannot say definitely which components of the program had impact, only that as a whole the investigators did see improvements.

In light of the above evidence regarding physical activity's impact on well being, one could reasonably offer that as a society we have a moral and ethical obligation to promote physical activity as a first-line treatment for depression. The question remains 'how can individuals, dealing with depression, be better motivated to become more physically active?' The promotion of physical activity through GMVs and the inclusion of a physical activity component within group patient visits are worthy of further investigation.

STUDY PROPOSAL: Through a mixed methods approach the investigators will evaluate the success of Jump Step, a series of 14 Group Medical Visits in motivating adults (≥18yrs), dealing with depression to become more physically active.

HYPOTHESIS: The investigators propose that adults dealing with Major Depressive Disorder (MDD) and/or Bi Polar II, depression, who participate in a weekly series of 14 Group Medical Visits (Jump Step) will have lower depression and anxiety ratings, higher rates of physical activity/step counts, and higher levels of "patient activation" post-intervention as compared to pre-intervention. Participants will also report deeper engagement and confidence in physical activity; increased levels of self-care and treatment as well as greater well being in qualitative interviews.

The investigators will recruit volunteers via the following approaches:

1. Posters located in A) the Mood Disorders Association of BC (MDABC); B) the psychiatric services area of major hospitals; C) areas visible to potential volunteers within related services organizations; D) coffee shops, community centres, YMCAs, and such venues. The investigators will obtain permission from the appropriate authorities to display advertisements;
2. Postings on the websites/list-serves of related service organizations such as the MDABC, the BC Psychiatric Association, BC Mental Health & Addiction Services, and Health Authority Mental Health Services. The investigators will obtain permission from the appropriate authorities to display advertisements;
3. Through word-of-mouth at MDABC and other service agencies and any resulting 'snowball sampling'.
4. Through social media such as Facebook and Twitter.
5. If needed the investigators will advertise in Lower Mainland papers.

MDABC psychiatrists and staff will also verbally inform clients of the opportunity to participate with the understanding that participation or non-participation will not affect a client's access to or quality of psychiatric care and/or MDABC services.

Previous participants in the Jump Step Needs Assessment (Part 1) (UBC Ethics: H14-00973) who meet the eligibility criteria and have signed consent will be given first preference.

Volunteers will either be emailed a blank consent form and a Physical Activity Readiness Questionnaire (2014 PAR-Q+) or obtain them through the MDABC office. Potential participants will scan and email their signed consent form and the PARQ+ form and Participant Declaration back to the Research Assistant; or they will mail signed paper copies of the forms back to the office of the investigators at the CHHM. Self Addressed Stamped Envelopes (SASEs) will be available at the MDABC office for this purposed. If needed the investigators will mail consent forms to potential participant along with a SASE.

Participants will have up to one-week prior to the baseline assessment or a minimum of 48 hours to review the consent form, ask questions, and/or discuss the consent with family members, friends, etc. The investigators believe 48 hours provides sufficient time for reflection and/or conversation and provides their Research Assistant with sufficient time to adequate schedule interviews.

Potential participants will contact their Research Assistant who will answer questions, confirm their eligibility, and schedule them for interviews. Each potential participant will have filled out, signed, and submitted the Physical Activity Readiness Questionnaire (2014 PAR-Q+). Research staff and/or the psychiatrist will follow up as appropriate, regarding their responses in the PARQ+.

Each assessment (baseline/post-intervention) will take approximately 90 minutes. The investigators will reimburse each participant $5 for each assessment they attend as well their parking/public transit up to $5.50 per assessment.

Professional transcription services will transcribe the interviews. Jump Step investigators will then analyze the data for common themes.

Intervention participants who have signed consent will be divided into cohorts of 20 participants each. Cohorts will participate in a weekly series of 14 Group Medical Visits (GMVs) co-led by a MDABC psychiatrist and an exercise therapist. GMVs will take place at the centrally located Robert Lee YMCA (downtown Vancouver), which will provide access to both meeting space for the group discussions as well as exercise facilities for the physical activity component of each Visit.

The curriculum will include (i) life skills development; (ii) disease specific education, relating to physical activity promotion, uptake, and adherence. The investigators will present also this education within a broader holistic context that acknowledges and supports a participant's social, emotional, spiritual, financial, physical, and nutritional well being; and (iii) GMVs will integrate medical care/medication management into their delivery.

During the physical activity component, participants will take part in regular group walks, emphasizing that 150 minutes weekly of moderate activity (e.g. brisk walking) is all that is necessary to obtain the medical benefits offered by regular physical activity. On other weeks participants will stay in the YMCA and be taught techniques and exercises that they can employ in their everyday lives to become more physically active without having to attend special classes, set aside time, or make concerted efforts to "exercise".

Group exercises might include aerobic training of cardio respiratory functioning, circuit training with simple tasks, e.g. ergometer bicycling, resistance bands, light weightlifting, etc. A trainer will supervise all interventions. Each subject will be given a physical activity sensor (Fit Bit) and participants will receive instruction from a researcher as to logging the wear time daily.

ELIGIBILITY:
We will recruit up to 80 participants who

Inclusion Criteria:

* are adults (≥18yrs)
* have a confirmed psychiatric assessment of Major Depressive Disorder (MDD) and/or Bipolar II, depressive
* are of moderate or higher severity (PHQ-9 >14)
* are community-dwelling and able to attend Group Medical Visits in the Lower Mainland
* are able to comply with scheduled visits, treatment plan, and other procedures;
* read, write, and speak English with acceptable auditory and visual acuity
* provide signed/dated informed consent; and
* able to walk independently.

Exclusion Criteria:

* Active psychotic symptoms
* a primary active diagnosis of substance abuse.

Participants will need to have a working proficiency in English as group discussions, accompanying texts, and instructions will all be in English. To provide adequate translation services for these elements in one or more other languages is beyond our budget and may also influence the dynamics of the GMV. It could be considered in a future iteration of this research program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
'Jump Step Intervention Questionnaire' | Post-Intervention (14 weeks)
  We will interview participants about physical activity levels, as well as their experience within the Jump Step intervention and its impact on their lives. We will also collect demographic data (age, gender, annual income, education level, self-identified disabilities, etc.)

SECONDARY OUTCOMES:
Physical Activity | Baseline
  We will measure participants' physical activity level (Actigraph; accelerometer).
Physical Activity | Post-Intervention (14 weeks)
  We will measure participants' physical activity level (Actigraph; accelerometer).
Patient Activation | Baseline
  a participants' levels of 'activation'
Patient Activation | Post-Intervention (14 weeks)
  a participants' levels of 'activation'
Anxiety | Baseline
  We will assess participants' anxiety ratings (GAD-7)
Anxiety | Post-Intervention (14 weeks)
  We will assess participants' anxiety ratings (GAD-7)
Social Support | Baseline
  We will assess participants' levels of social support (abridged Berlin Social Support Scales (BSSS))
Social Support | Post-Intervention (14 weeks)
  We will assess participants' levels of social support (abridged Berlin Social Support Scales (BSSS))
Depression | Baseline
  We will assess participants' depression ratings via the PHQ-9.
Depression | Post-Intervention (14 weeks)
  We will assess participants' depression ratings via the PHQ-9.

OTHER OUTCOMES:
'Jump Step Facilitators Questionnaire' | Baseline
  We will interview the Jump Step facilitators about their experience of the intervention.
'Jump Step Facilitators Questionnaire' | Post-Intervention (14 weeks)
  We will interview the Jump Step facilitators about their experience of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Joanie Sims-Gould, PhD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Centre for Hip Health & Mobility, Department of Family Practice, Vancouver, British Columbia
  - Mood Disorders Association of BC, Vancouver, British Columbia
  - Robert Lee YMCA, Vancouver, British Columbia